CLINICAL TRIAL: NCT06901037
Title: The Acceptability and Preliminary Effectiveness of Using A Smartphone-delivered AI-Based Chatbot in Older Adults for Lifestyle Modification: A Pilot Randomized Controlled Trial
Brief Title: A Pilot Randomized Controlled Trial of Chatbot Use in Older Adults for Lifestyle Change
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Associate Professor in the School of Nursing, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSEARS20250305010
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Healthy Lifestyle
Keywords: Chatbot, older adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot-based intervention (Experimental): Participants will immediately receive access to a 2-month chatbot-based intervention
  Interventions: Other: A chatbot-based intervention
- Waitlist (Other): Participants will be placed on a waiting list before accessing the intervention
  Interventions: Other: A chatbot-based intervention

INTERVENTIONS:
Other: A chatbot-based intervention — A smartphone-delivered AI-based chatbot program designed to provide personalized physical activity and dietary recommendations

SUMMARY:
The purpose of this study is to evaluate the acceptability and preliminary effectiveness of a smartphone-delivered AI-based chatbot in promoting healthy dietary behavior and physical activity participation among older adults.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the preliminary effectiveness of a smartphone-delivered AI-based chatbot in promoting healthy dietary behavior and physical activity participation among older adults. It is a preliminary study with two arms.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or above.
* are community-dwelling.
* are proficient in Mandarin.
* have an Internet connection.
* have at least one instant messaging app on the smartphone or agree to download one.

Exclusion Criteria:

* have any neurocognitive disorders.
* are unable to engage in moderate-intensity level of physical activity due to a preexisting medical condition.
* live with another participant who will participate in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The acceptance of the chatbot among older adults, as measured by a 14-item simplified version of the Senior Technology Acceptance Model questionnaire | End of study (2 months)
  The 14-item questionnaire uses a 10-point Likert scale, ranging from 0 (strongly disagree, very poor, very uneasy, and very unsatisfied) to 10 (strongly agree, very good, very easy, and very satisfied)
The Usability of the chatbot, as measured by the System Usability Scale | End of study (2 months)
  The System Usability Scale (SUS) is a 10-item Likert scale questionnaire. The result of this survey is called SUS score, which ranges from 0 to 100 and provides information about overall customer satisfaction and usability. A higher score indicates better usability, while a lower score may suggest usability issues.
The user experience, as measured by 10 open-ended questions | End of study (2 months)
  A qualitative interview will be provided to the participants for asking their experience in using chatbot.

SECONDARY OUTCOMES:
Change of dietary behavior, as measured by the intake of fruits and vegetables over the last seven days | Baseline, end of study (2 months)
  We will ask them the amount of fruit and vegetable intake at baseline and end of study.
Change of walking, as measured by the Community Health Activities Model Program for Seniors questionnaire | Baseline, end of study (2 months)
  The Community Health Activities Model Program for Seniors questionnaires (CHAMPS-Q) measures weekly frequency and duration of walking
Change of total activity and moderate and more vigorous physical activity variables, as measured by the CHAMPS-Q | Baseline, end of study (2 months)
  The CHAMPS-Q measures weekly frequency and duration of a variety of lifestyle physical activities
Change of quality of life, as measured by the Hong Kong Quality of Life for Older Persons Scale | Baseline, end of study (2 months)
  The Hong Kong Quality of Life for Older Persons Scale (HKQoLOCP) comprises a total of 21 items that can be categorized into different domains: subjective well-being, consisting of 4 items; health, comprising 5 items; interpersonal relationships, including 6 items; achievement-recognition, with 4 items; and finance and living conditions (1 item each)

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No sharing of data except reasonable request.